CLINICAL TRIAL: NCT05524012
Title: Planning Adaptive Treatment by Longitudinal Response Assessment Implementing MR Imaging, Liquid Biopsy and Analysis of Microenvironment During Neoadjuvant Treatment of Rectal Cancer (PRIMO)
Brief Title: Longitudinal Multimodal Response Assessment During Neoadjuvant Treatment of Rectal Cancer
Acronym: PRIMO
Status: Active, not recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Georg Wurschi, Principal Investigator, Jena University Hospital
Other Study IDs: UKJ-PRIMO-2022; CSP-11 (Other Grant/Funding Number: Clinician Scientist Program, Interdisciplinary Center for Clinical Research, Jena University Hospital); LIFE Talent Funds 2022 (Other Grant/Funding Number: Friedrich Schiller University)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Rectal Carcinoma; Neoadjuvant Treatment; Radiotherapy; Adaptive Treatment
Keywords: total neoadjuvant therapy (TNT); T2* MRI; circulating tumor cells; tumor infiltrating lymphocytes; liquid biopsy; DWI; rectal cancer; organ preservation
MeSH Terms: conditions — Neoplastic Cells, Circulating; Rectal Neoplasms | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * histological analysis of tumor specimens (pre-treatment biopsy and resected tumor)
  * blood samples (Circulating Tumor Cells, CTCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood sample — longitudinal blood samples for CTC monitoring
  Other Names: analyses of circulating tumor cells (CTC)
Device: MRI scan — longitudinal MRI scans (non-contrast enhanced)
  Other Names: multiparametric (incl. DWI and T2* "BOLD")

SUMMARY:
This pilot study aims to trial multimodal early response assessment to enable therapy adaptions in the context of non-operative therapy strategies of locally advanced rectal cancer (LARC) for development of a non-invasive response prediction model.

DETAILED DESCRIPTION:
Patients with LARC, receiving neoadjuvant chemoradiotherapy (CRT) are followed by at least 4 multiparametric MRI-scans (diffusion weighted imaging and hypoxia-sensitive sequences) as well as repeated blood samples in order to analyse circulating tumour cells (CTCs). A standard pelvis radiotherapy (RT, 5040 cGy) will be performed in combination with a 5-Fluorouracil / Oxaliplatin regimen in all patients (planned: N = 50), succeeded by consolidation CTx (FOLFOX4) if feasible. Additional histologic markers, such as tumour-infiltrating lymphocytes (TILs) or PD-L1 status will be analysed before and after CRT. Resection is standard after completion of preoperative treatment. In case of complete regression and patient's request, a non-operative management ("watch and wait") is offered alternatively. The primary endpoint is response, defined by tumor regression grading, secondary endpoints comprise longitudinal changes in MRI as well as in CTCs and TILs.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced rectal cancer (LARC): UICC Stage II/III
* no severe cardiac or lung disease
* no severe hepatic disorders (liver enzymes <2.5 NR) or restrictions of renal function (GFR > 30ml/min)
* no severe cytopenia (Neutrocytes >= 3 Gpt/l; Thrombocytes >= 100 Gpt/l; Hemoglobin >6mmol/l)
* no homozygotic DPD deficiency
* no other neoplasms requiring therapy
* no earlier radiotherapy of the pelvis or earlier chemotherapy
* no contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer (LARC), receiving neoadjuvant chemoradiotherapy (CRT).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Tumor regression grading (TRG) | after completion of neoadjuvant treatment (up to 10 months)
  Histological response assessment by TRG (Werner / Hoefler et al.); Complete response is defined as TRG 1a;

SECONDARY OUTCOMES:
MRI | up to 10 months, until resection
  longitudinal changes in multiparametric MRI sequences (diffusion weighted and hypoxia sensitive)
Circulating Tumor Cells (CTC) | 5 years
  longitudinal changes in CTCs
Tumor Infiltrating Lymphocytes (TIL) | up to 10 months, until resection
  longitudinal changes in TILs
PFS | 5 years
  progression free survival
OS | 5 years
  overall survival
Surrogate marker: Interleukin 6 (IL-6) | 5 years
  surrogates of tumor and inflammation from routine blood draws [ng/l]
Surrogate marker: Carcinoembryonic Antigen (CEA) | 5 years
  surrogates of tumor and inflammation from routine blood draws, [mg/l]

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wittig-Sauerwein, MD, Principal Investigator — Department for Radiotherapy and Radiooncology, Jena University Hospital
Locations (1):
- Department of Radiotherapy and Radiation Oncology, Jena University Hospital, Jena, Germany

IPD SHARING:
Plan to Share IPD: No